Protocol 17-24231 Confidential

## JOHN V. FAHY, MD, MSC Clinical Research Protocol INPATIENT CLINICAL TRIAL OF NAC IN ASTHMA (ICON)

| Protocol Number: | 17-24231 |
|--------------------------|--------------------------------|
| NCT Number | NCT03581084 |
| Investigational Product: | n-acetylcysteine |
| Development Phase: | 4 |
| Sponsor: | John V. Fahy, MD, MSc |
| | 513 Parnassus Avenue, HSE 1307 |
| | San Francisco, CA 94143-0130 |
| Funding Organization: | NIH |
| Principal Investigator: | Name: John V. Fahy, MD, MSc |
| | Telephone: 415-476-9940 |
| | Fax: 415-476-5712 |
| | E-mail: John.Fahy@ucsf.edu |

## STATISTICAL ANALYSIS PLAN

Our overarching method (experimental approach) is to test the efficacy of inhaled NAC delivered for 5 days to asthma patients who have baseline evidence of mucus plugs on CT lung scans. We will assess if the NAC treatment causes the mucus plugs to go away by the end of the treatment period and we will assess for reappearance of mucus plugs at 6 weeks and 3 months time. We will also examine whether any NAC associated decrease in mucus plugs is associated with improvement in FEV1. A primary analysis will be paired T-test analysis of the change in CT mucus plug score and in FEV1 from baseline to end treatment. Secondary analyses will look at the 6 week and 3 month time points.

Version 11/8/2018